CLINICAL TRIAL: NCT01251653
Title: A Phase I Dose Escalation Trial of Once Daily Oral Treatment Using Afatinib (BIBW2992) Plus Gemcitabine or Docetaxel in Patients With Relapsed or Refractory Solid Tumors.
Brief Title: A Phase I Dose Escalation Trial of Afatinib Plus Gemcitabine or Plus Docetaxel
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1200.93; 2010-020560-37 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-04

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Afatinib; Docetaxel; Gemcitabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Pharmacokinetic samples

GROUPS / COHORTS (2):
- Afatinib and docetaxel
  Interventions: Drug: Afatinib; Drug: docetaxel
- Afatinib and gemcitabine
  Interventions: Drug: Afatinib; Drug: gemcitabine

INTERVENTIONS:
Drug: Afatinib — Maximum Tolerated Dose of Afatinib in combination with gemcitabine
  Groups: Afatinib and docetaxel
Drug: Afatinib — Maximum Tolerated Dose of Afatinib in combination with gemcitabine
  Groups: Afatinib and gemcitabine
Drug: docetaxel — Maximum Tolerated Dose of Afatinib in combination with docetaxel
  Groups: Afatinib and docetaxel
Drug: gemcitabine — Maximum Tolerated Dose of Afatinib in combination with gemcitabine
  Groups: Afatinib and gemcitabine

SUMMARY:
To establish the maximum tolerated dose (MTD) of oral afatinib (BIBW2992) given in combination with gemcitabine or docetaxel in patients with relapsed or refractory tumors.

To assess the safety of the combination. To investigate the PK characteristics of docetaxel or gemcitabine and of oral afatinib (BIBW2992) in the tested treatment schedule. To assess antitumor activity.

ELIGIBILITY:
Inclusion criteria:

1. histologically or cytologically confirmed diagnosis of any advanced or metastatic relapsed or refractory solid tumor.

Exclusion criteria:

1. Active brain metastases
2. Patients with known pre-existing interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: solid tumors
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2010-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (3):
- France (3):
  - 1200.93.33002 Boehringer Ingelheim Investigational Site, Dijon
  - 1200.93.33001 Boehringer Ingelheim Investigational Site, Saint-Herblain
  - 1200.93.33003 Boehringer Ingelheim Investigational Site, Toulouse

REFERENCES:
- [Derived] Hiret S, Isambert N, Gomez-Roca C, Bennouna J, Sassi M, de Mont-Serrat H, Fan J, Schnell D, Delord JP. Phase I dose-escalation trial of afatinib, an irreversible ErbB family blocker, in combination with gemcitabine or docetaxel in patients with relapsed or refractory solid tumors. Invest New Drugs. 2018 Dec;36(6):1044-1059. doi: 10.1007/s10637-018-0601-1. Epub 2018 May 29. PMID 29808308

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were completed the study but discontinued from the trial medication
Pre-assignment Details: This was an uncontrolled, open-label, Phase I, '3+3' dose-escalation trial to determine the maximum tolerated dose (MTDs) for combination Afatinib with Gemcitabine or with Docetaxel; 2 MTDs were to be defined, one for Afatinib with Gemcitabine (Cohort A) and one for Afatinib with Docetaxel (Cohort B).
Groups:
- Afatinib 30mg and Gemcitabine 1000mg: Afatinib (film-coated tablet) 30 mg qd (once daily) was administered orally in combination with Gemcitabine 1000 mg/m2 administered as intravenous infusion on Days 1 and 8 of each 3- week treatment course.
- Afatinib 30mg and Gemcitabine 1250mg: Afatinib (film-coated tablet) 30 mg qd (once daily) was administered orally in combination with Gemcitabine 1250 mg/m2 administered as intravenous infusion on Days 1 and 8 of each 3- week treatment course.
- Afatinib 40mg and Gemcitabine 1000mg: Afatinib (film-coated tablet) 40 mg qd (once daily) was administered orally in combination with Gemcitabine 1000 mg/m2 administered as intravenous infusion on Days 1 and 8 of each 3- week treatment course.
- Afatinib 40mg and Gemcitabine 1250mg: Afatinib (film-coated tablet) 40 mg qd (once daily) was administered orally in combination with Gemcitabine 1250 mg/m2 administered as intravenous infusion on Days 1 and 8 of each 3- week treatment course.
- Afatinib 50mg and Gemcitabine 1250mg: Afatinib (film-coated tablet) 50 mg qd (once daily) was administered orally in combination with Gemcitabine 1250 mg/m2 administered as intravenous infusion on Days 1 and 8 of each 3- week treatment course.
- Afatinib 30mg and Docetaxel 60mg: Afatinib (film-coated tablet) 30 mg qd (once daily) was administered orally in combination with Docetaxel 60 mg/m2 administered as intravenous infusion on Day 1 of each 3- week treatment course
- Afatinib 30mg and Docetaxel 75mg: Afatinib (film-coated tablet) 30 mg qd (once daily) was administered orally in combination with Docetaxel 75 mg/m2 administered as intravenous infusion on Day 1 of each 3- week treatment course.
- Afatinib 40mg and Docetaxel 75mg: Afatinib (film-coated tablet) 40 mg qd (once daily) was administered orally in combination with Docetaxel 75 mg/m2 administered as intravenous infusion on Day 1 of each 3- week treatment course.
- Afatinib 50mg and Docetaxel 75mg: Afatinib (film-coated tablet) 50 mg qd (once daily) was administered orally in combination with Docetaxel 75 mg/m2 administered as intravenous infusion on Day 1 of each 3- week treatment course.
Period: Overall Study
Arm/Group | Afatinib 30mg and Gemcitabine 1000mg | Afatinib 30mg and Gemcitabine 1250mg | Afatinib 40mg and Gemcitabine 1000mg | Afatinib 40mg and Gemcitabine 1250mg | Afatinib 50mg and Gemcitabine 1250mg | Afatinib 30mg and Docetaxel 60mg | Afatinib 30mg and Docetaxel 75mg | Afatinib 40mg and Docetaxel 75mg | Afatinib 50mg and Docetaxel 75mg
Started | 3 | 8 | 20 | 6 | 2 | 18 | 18 | 12 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 8 | 20 | 6 | 2 | 18 | 18 | 12 | 6
Not completed — Progressive Disease | 1 | 7 | 16 | 4 | 0 | 17 | 14 | 7 | 5
Not completed — Dose-limiting toxicity | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 2 | 1 | 1 | 0 | 2 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Other reason not mentioned above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): The Treated Set consists of all patients who received at least one application of the trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Afatinib 30mg and Gemcitabine 1000mg | Afatinib 30mg and Gemcitabine 1250mg | Afatinib 40mg and Gemcitabine 1000mg | Afatinib 40mg and Gemcitabine 1250mg | Afatinib 50mg and Gemcitabine 1250mg | Afatinib 30mg and Docetaxel 60mg | Afatinib 30mg and Docetaxel 75mg | Afatinib 40mg and Docetaxel 75mg | Afatinib 50mg and Docetaxel 75mg | Total
Number analyzed (Participants) | 3 | 8 | 20 | 6 | 2 | 18 | 18 | 12 | 6 | 93
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.7 (20.8) | 52.1 (13.8) | 57.7 (10.2) | 52.3 (16.5) | 61.0 (1.4) | 55.4 (11.0) | 59.2 (10.6) | 59.3 (10.2) | 54.5 (6.5) | 56.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 10 | 5 | 1 | 9 | 10 | 5 | 3 | 49
  Male | 2 | 3 | 10 | 1 | 1 | 9 | 8 | 7 | 3 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) in Process for the Determination of the Maximum Tolerated Dose (MTD).
Description: DLT was based on following criterions: 1. Grade 4 uncomplicated (not associated with fever >38.5° C (Celsius)) neutropenia for ≥7 days. 2. Grade 3 or 4 neutropenia concomitant with fever >38.5º C or Grade ≥3 infection. 3. Platelet count of <25x 10^9/L or <50x 10^9/L with bleeding requiring whole blood transfusion. 4. Grade ≥3 non-haematological toxicity (except untreated nausea, untreated vomiting, or untreated diarrhoea). 5. Grade ≥2 decrease in cardiac left ventricular function. 6. Grade ≥2 worsening of renal function as measured by serum creatinine, newly developed proteinuria, or a newly developed decrease in glomerular filtration rate. Toxicity grading was based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3.0
Time Frame: 3 weeks
Population: Treated Set (TS)
Measure: Number; unit: Participants
Arm/Group | Afatinib 30mg and Gemcitabine 1000mg | Afatinib 30mg and Gemcitabine 1250mg | Afatinib 40mg and Gemcitabine 1000mg | Afatinib 40mg and Gemcitabine 1250mg | Afatinib 50mg and Gemcitabine 1250mg | Afatinib 30mg and Docetaxel 60mg | Afatinib 30mg and Docetaxel 75mg | Afatinib 40mg and Docetaxel 75mg | Afatinib 50mg and Docetaxel 75mg
Number analyzed (Participants) | 3 | 8 | 20 | 6 | 2 | 18 | 18 | 12 | 6
Participants | 0 | 1 | 1 | 2 | 2 | 4 | 6 | 5 | 1

2. Secondary Outcome: The Incidence and Intensity of AEs With Grading According to CTCAE.
Description: The incidence and intensity of adverse events with grading according to CTCAE. The CTCAE grades are: 1 (mild AE), 2 (moderate AE), 3 (severe AE), 4 (life-threatening or disabling AE), 5 (death related to AE).
Time Frame: From first drug administration until 28 days after last drug administration, up to 717 days.
Population: TS
Measure: Number; unit: Participants
Arm/Group | Afatinib 30mg and Gemcitabine 1000mg | Afatinib 30mg and Gemcitabine 1250mg | Afatinib 40mg and Gemcitabine 1000mg | Afatinib 40mg and Gemcitabine 1250mg | Afatinib 50mg and Gemcitabine 1250mg | Afatinib 30mg and Docetaxel 60mg | Afatinib 30mg and Docetaxel 75mg | Afatinib 40mg and Docetaxel 75mg | Afatinib 50mg and Docetaxel 75mg
Number analyzed (Participants) | 3 | 8 | 20 | 6 | 2 | 18 | 18 | 12 | 6
Participants
  Grade 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 | 2 | 1 | 5 | 2 | 0 | 3 | 1 | 0 | 1
  Grade 3 | 0 | 6 | 6 | 2 | 1 | 6 | 4 | 4 | 2
  Grade 4 | 0 | 1 | 5 | 1 | 1 | 6 | 11 | 6 | 1
  Grade 5 | 1 | 0 | 4 | 1 | 0 | 2 | 2 | 2 | 2

3. Secondary Outcome: Best Overall Response According to RECIST v1.1 Criteria
Description: Best overall response (according to Response Evaluation Criteria in Solid Tumours [RECIST] version 1.1) was the best response recorded at any time from the date of the first administration of afatinib or gemcitabine/docetaxel to the end of treatment (EOT). Partial response is for patients with measurable disease. Missing categories signifies that no tumour imaging has been performed post baseline, and therefore the response status could not be assessed.
Time Frame: From first drug administration until 28 days after last drug administration, up to 717 days.
Population: TS
Measure: Number; unit: Participants
Arm/Group | Afatinib 30mg and Gemcitabine 1000mg | Afatinib 30mg and Gemcitabine 1250mg | Afatinib 40mg and Gemcitabine 1000mg | Afatinib 40mg and Gemcitabine 1250mg | Afatinib 50mg and Gemcitabine 1250mg | Afatinib 30mg and Docetaxel 60mg | Afatinib 30mg and Docetaxel 75mg | Afatinib 40mg and Docetaxel 75mg | Afatinib 50mg and Docetaxel 75mg
Number analyzed (Participants) | 3 | 8 | 20 | 6 | 2 | 18 | 18 | 12 | 6
Participants
  Complete response (CR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial response | 0 | 1 | 4 | 0 | 0 | 1 | 5 | 4 | 0
  Stable disease/ Non-CR/Non-PD | 2 | 3 | 9 | 5 | 0 | 9 | 8 | 5 | 2
  Progressive disease (PD) | 1 | 3 | 6 | 1 | 2 | 8 | 4 | 2 | 4
  Not evaluable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Missing | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0

4. Secondary Outcome: Disease Control According to RECIST v1.1
Description: Disease control according to RECIST v1.1 Disease control is complete response, partial response or stable disease for measurable patients and complete response or non-CR/non-PD for non-measurable patients. Missing categories signify that no tumour imaging has been performed post baseline, and therefore the response status could not be assessed.
Time Frame: From first drug administration until 28 days after last drug administration, up to 717 days.
Population: TS
Measure: Number; unit: Participants
Arm/Group | Afatinib 30mg and Gemcitabine 1000mg | Afatinib 30mg and Gemcitabine 1250mg | Afatinib 40mg and Gemcitabine 1000mg | Afatinib 40mg and Gemcitabine 1250mg | Afatinib 50mg and Gemcitabine 1250mg | Afatinib 30mg and Docetaxel 60mg | Afatinib 30mg and Docetaxel 75mg | Afatinib 40mg and Docetaxel 75mg | Afatinib 50mg and Docetaxel 75mg
Number analyzed (Participants) | 3 | 8 | 20 | 6 | 2 | 18 | 18 | 12 | 6
Participants
  No | 1 | 3 | 6 | 1 | 2 | 8 | 4 | 2 | 4
  Yes | 2 | 4 | 13 | 5 | 0 | 10 | 13 | 9 | 2
  Missing | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0

5. Secondary Outcome: Objective Response According to RECIST v1.1
Description: Objective response according to RECIST v1.1. Objective response is complete response or partial response for patients with measurable disease. Missing categories signify that no tumour imaging has been performed post baseline, and therefore the response status could not be assessed.
Time Frame: From first drug administration until 28 days after last drug administration, up to 717 days.
Population: TS
Measure: Number; unit: Participants
Arm/Group | Afatinib 30mg and Gemcitabine 1000mg | Afatinib 30mg and Gemcitabine 1250mg | Afatinib 40mg and Gemcitabine 1000mg | Afatinib 40mg and Gemcitabine 1250mg | Afatinib 50mg and Gemcitabine 1250mg | Afatinib 30mg and Docetaxel 60mg | Afatinib 30mg and Docetaxel 75mg | Afatinib 40mg and Docetaxel 75mg | Afatinib 50mg and Docetaxel 75mg
Number analyzed (Participants) | 3 | 8 | 20 | 6 | 2 | 18 | 18 | 12 | 6
Participants
  No | 3 | 6 | 15 | 6 | 2 | 17 | 12 | 7 | 6
  Yes | 0 | 1 | 4 | 0 | 0 | 1 | 5 | 4 | 0
  Missing | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0

6. Secondary Outcome: Time to Objective Response According to RECIST v1.1
Description: Objective response according to RECIST v1.1. Objective response is complete response or partial response for patients with measurable disease. Time to objective response is the time from the start of treatment to the date of first documented complete response or partial response. Descriptive analyses has been performed for the time to objective response (N(%) of patients with first occurrence of objective response at 6, 12 and 24 weeks). Onset of objective response is derived for patient with measurable disease.
Time Frame: 6 weeks, 12 weeks and 24 weeks
Population: TS
Measure: Number; unit: Participants
Arm/Group | Afatinib 30mg and Gemcitabine 1000mg | Afatinib 30mg and Gemcitabine 1250mg | Afatinib 40mg and Gemcitabine 1000mg | Afatinib 40mg and Gemcitabine 1250mg | Afatinib 50mg and Gemcitabine 1250mg | Afatinib 30mg and Docetaxel 60mg | Afatinib 30mg and Docetaxel 75mg | Afatinib 40mg and Docetaxel 75mg | Afatinib 50mg and Docetaxel 75mg
Number analyzed (Participants) | 3 | 8 | 20 | 6 | 2 | 18 | 18 | 12 | 6
Participants
  6 Weeks | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 1 | 0
  12 Weeks | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 2 | 0
  24 Weeks | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Not applicable | 3 | 7 | 16 | 6 | 2 | 17 | 13 | 8 | 6

7. Secondary Outcome: Duration of Objective Response According to RECIST v1.1
Description: Duration of objective response was the time from the first documented complete response or partial response to disease progression or death.
Time Frame: From the first documented complete response or partial response to the time of disease progression or death
Population: TS for patients who experienced objective response.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Afatinib 30mg and Gemcitabine 1000mg | Afatinib 30mg and Gemcitabine 1250mg | Afatinib 40mg and Gemcitabine 1000mg | Afatinib 40mg and Gemcitabine 1250mg | Afatinib 50mg and Gemcitabine 1250mg | Afatinib 30mg and Docetaxel 60mg | Afatinib 30mg and Docetaxel 75mg | Afatinib 40mg and Docetaxel 75mg | Afatinib 50mg and Docetaxel 75mg
Number analyzed (Participants) | 0 | 1 | 4 | 0 | 0 | 1 | 5 | 4 | 0
Days |  | 291.0 (NA) — Non Calculable as only one participant analysed. | 138.3 (80.2) |  |  | 410.0 (NA) — Non Calculable as only one participant analysed. | 296.0 (132.8) | 55.5 (64.4) |

8. Secondary Outcome: Duration of Disease Control According to RECIST v1.1
Description: Duration of disease control according to RECIST v1.1.
Time Frame: From the first administration of study medication to the time of disease progression or death
Population: TS for patients who experienced disease control.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Afatinib 30mg and Gemcitabine 1000mg | Afatinib 30mg and Gemcitabine 1250mg | Afatinib 40mg and Gemcitabine 1000mg | Afatinib 40mg and Gemcitabine 1250mg | Afatinib 50mg and Gemcitabine 1250mg | Afatinib 30mg and Docetaxel 60mg | Afatinib 30mg and Docetaxel 75mg | Afatinib 40mg and Docetaxel 75mg | Afatinib 50mg and Docetaxel 75mg
Number analyzed (Participants) | 2 | 4 | 13 | 5 | 0 | 10 | 13 | 9 | 2
Days | 119.5 (68.6) | 210.0 (118.1) | 119.7 (148.5) | 77.4 (19.9) |  | 207.1 (108.1) | 233.6 (150.8) | 158.7 (89.0) | 85.0 (8.5)

9. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival was defined as the time from the first administration of study medication to the time of disease progression or death, whichever occurred first.
Time Frame: From the first administration of study medication to the time of disease progression or death
Population: TS, MTD cohort
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Afatinib 40mg and Gemcitabine 1000mg | Afatinib 30mg and Docetaxel 60mg | Afatinib 30mg and Docetaxel 75mg
Number analyzed (Participants) | 20 | 18 | 18
Weeks | 23.9 (148.5) [5.9 to 25.0] | 18.1 (108.1) [5.7 to 31.3] | 23.6 (150.8) [7.0 to 31.6]

10. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from the first administration of study medication to the time of death from any cause.
Time Frame: From the first administration of study medication to the time of death
Population: TS, MTD cohort
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Afatinib 40mg and Gemcitabine 1000mg | Afatinib 30mg and Docetaxel 60mg | Afatinib 30mg and Docetaxel 75mg
Number analyzed (Participants) | 20 | 18 | 18
Weeks | 52.4 (148.5) [35.4 to NA] — Non calculable because the 75th percentile hasn't been reached | 38.4 (108.1) [26.0 to NA] — Non calculable because the 75th percentile hasn't been reached | NA (150.8) [68.1 to NA] — Non calculable because the median hasn't been reached

11. Secondary Outcome: Area Under the Concentration-time Curve (AUC) Tau,ss of Afatinib
Description: Area under the concentration-time curve of Afatinib in plasma over a uniform dosing interval t at steady state.
Time Frame: PK samples were taken at hours; 167:55, 479:55, 481:05, 482:05, 483:05, 485:05, 487:05 and on day 22 at hours; -0:10, 1, 2, 3, 5, 7, 23:55
Population: The Pharmacokinetic Set (PKS) was a subset of the Treated Set that included all patients who had taken at least 1 dose of study medication and for whom at least 1 valid plasma concentration was available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Afatinib 40mg With Gemcitabine 1000 mg: Afatinib (film-coated tablet) 40 mg qd (once daily) was administered orally in combination with Gemcitabine 1000 mg/m2 administered as intravenous infusion on Days 1 and 8 of each 3- week treatment course.
- Afatinib 40mg Without Gemcitabine: Afatinib (film-coated tablet) 40 mg qd (once daily) was administered orally in 3- week treatment course.
- Afatinib 30mg With Docetaxel 60mg: Afatinib (film-coated tablet) 30 mg qd (once daily) was administered orally in combination with Docetaxel 60 mg/m2 administered as intravenous infusion on Day 1 of each 3- week treatment course
- Afatinib 30mg Without Docetaxel 60mg; Afatinib 30mg Without Docetaxel 75mg: Afatinib (film-coated tablet) 30 mg qd (once daily) was administered orally in 3- week treatment course.
- Afatinib 30mg With Docetaxel 75mg: Afatinib (film-coated tablet) 30 mg qd (once daily) was administered orally in combination with Docetaxel 75 mg/m2 administered as intravenous infusion on Day 1 of each 3- week treatment course.
Arm/Group | Afatinib 40mg With Gemcitabine 1000 mg | Afatinib 40mg Without Gemcitabine | Afatinib 30mg With Docetaxel 60mg | Afatinib 30mg Without Docetaxel 60mg | Afatinib 30mg With Docetaxel 75mg | Afatinib 30mg Without Docetaxel 75mg
Number analyzed (Participants) | 8 | 5 | 12 | 12 | 14 | 10
ng*h/mL | 1000.0 (24.5) | 1230.0 (113.0) | 642.0 (64.0) | 746.0 (61.6) | 557.0 (54.0) | 723.0 (58.3)
Statistical Analysis 1: Comparison: Afatinib 40mg With Gemcitabine 1000 mg vs Afatinib 40mg Without Gemcitabine; Test type: Non-Inferiority or Equivalence — p-value for ratio outside interval 80% to 125%; p = 0.4815, ANOVA; ANOVA (analysis of variance) model on the logarithm scale was used with 'subject' as random, whereas the 'treatment' as fixed effect; Ratio of adjusted gmeans in percentage = 81.27, 90% CI 2-sided [44.863 to 147.205], Standard Deviation 63.3 — Relative bioavailability of Afatinib with Gemcitabine vs. Afatinib without Gemcitabine was estimated by the ratios of the adjusted geometric means (gMean). Standard deviation is actually intra-individual geometric coefficient variation (gCV)
Statistical Analysis 2: Comparison: Afatinib 30mg With Docetaxel 60mg vs Afatinib 30mg Without Docetaxel 60mg; Test type: Non-Inferiority or Equivalence — p-value for ratio outside interval 80% to 125%; p = 0.0149, ANOVA; [statistical method as in outcome 11, analysis 1]; Ratio of adjusted gmeans in percentage = 95.36, 90% CI 2-sided [84.139 to 108.077], Standard Deviation 15.4 — Relative bioavailability of Afatinib with Docetaxel vs. Afatinib without Docetaxel was estimated by the ratios of the adjusted geometric means (gMean). Standard deviation is actually intra-individual geometric coefficient variation (gCV)
Statistical Analysis 3: Comparison: Afatinib 30mg With Docetaxel 75mg vs Afatinib 30mg Without Docetaxel 75mg; Test type: Non-Inferiority or Equivalence — p-value for ratio outside interval 80% to 125%; p = 0.0208, ANOVA; [statistical method as in outcome 11, analysis 1]; Ratio of adjusted gmeans in percentage = 88.12, 90% CI 2-sided [81.778 to 94.964], Standard Deviation 9.2 — [estimate comment as in outcome 11, analysis 2]

12. Secondary Outcome: Cmax,ss of Afatinib
Description: Maximum concentration of Afatinib in plasma at steady state.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Afatinib 40mg With Gemcitabine 1000 mg | Afatinib 40mg Without Gemcitabine | Afatinib 30mg With Docetaxel 60mg | Afatinib 30mg Without Docetaxel 60mg | Afatinib 30mg With Docetaxel 75mg | Afatinib 30mg Without Docetaxel 75mg
Number analyzed (Participants) | 9 | 6 | 14 | 13 | 15 | 10
ng/mL | 58.1 (73.3) | 66.4 (106.0) | 33.9 (70.2) | 45.6 (78.7) | 33.9 (50.6) | 45.7 (68.3)
Statistical Analysis 1: Comparison: Afatinib 40mg With Gemcitabine 1000 mg vs Afatinib 40mg Without Gemcitabine; Test type: Non-Inferiority or Equivalence — p-value for ratio outside interval 80% to 125%; p = 0.8715, ANOVA; [statistical method as in outcome 11, analysis 1]; Ratio of adjusted gmeans in percentage = 141.36, 90% CI 2-sided [115.848 to 172.495], Standard Deviation 14.7 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Afatinib 30mg With Docetaxel 60mg vs Afatinib 30mg Without Docetaxel 60mg; Test type: Non-Inferiority or Equivalence — p-value for ratio outside interval 80% to 125%; p = 0.6805, ANOVA; [statistical method as in outcome 11, analysis 1]; Ratio of adjusted gmeans in percentage = 77.42, 90% CI 2-sided [68.516 to 87.473], Standard Deviation 16.8 — [estimate comment as in outcome 11, analysis 2]
Statistical Analysis 3: Comparison: Afatinib 30mg With Docetaxel 75mg vs Afatinib 30mg Without Docetaxel 75mg; Test type: Non-Inferiority or Equivalence — p-value for ratio outside interval 80% to 125%; p = 0.2327, ANOVA; [statistical method as in outcome 11, analysis 1]; Ratio of adjusted gmeans in percentage = 83.95, 90% CI 2-sided [74.794 to 94.217], Standard Deviation 14.3 — [estimate comment as in outcome 11, analysis 2]

13. Secondary Outcome: AUC 0-tz of Gemcitabine
Description: Area under the concentration-time curve of Gemcitabine in plasma over the time interval from 0 up to the last quantifiable data point
Time Frame: PK samples were taken on day 1 at hours; -0:05, 0:30, 1, 1:30, 2, 3 and on day 22 at hours; -0:10, 0:30, 1, 1:30, 2, 3
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Gemcitabine 1000mg With Afatinib 40 mg: Afatinib (film-coated tablet) 40 mg qd (once daily) was administered orally in combination with Gemcitabine 1000 mg/m2 administered as intravenous infusion on Days 1 and 8 of each 3- week treatment course.
- Gemcitabine 1000mg Without Afatinib: Gemcitabine 1000 mg/m2 administered as intravenous infusion on Days 1 and 8 of each 3- week treatment course.
Arm/Group | Gemcitabine 1000mg With Afatinib 40 mg | Gemcitabine 1000mg Without Afatinib
Number analyzed (Participants) | 11 | 13
ng*h/mL | 9610.0 (26.5) | 7120.0 (38.8)
Statistical Analysis 1: Comparison: Gemcitabine 1000mg With Afatinib 40 mg vs Gemcitabine 1000mg Without Afatinib; Test type: Non-Inferiority or Equivalence — p-value for ratio outside interval 80% to 125%; p = 0.7759, ANOVA; [statistical method as in outcome 11, analysis 1]; Ratio of adjusted gmeans in percentage = 136.11, 90% CI 2-sided [112.09 to 165.29], Standard Deviation 26.3 — Relative bioavailability of Gemcitabine with Afatinib vs. Gemcitabine without Afatinib was estimated by the ratios of the adjusted geometric means (gMean). Standard deviation is actually intra-individual geometric coefficient variation (gCV)

14. Secondary Outcome: Cmax of Gemcitabine
Description: Maximum concentration of Gemcitabine in plasma.
Time Frame: PK samples were taken on day 1 at hours; -0:05, 0:30, 1, 1:30, 2, 3 and on day 22 at hours; -0:10, 0:30, 1, 1:30, 2, 3
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Gemcitabine 1000mg With Afatinib 40 mg | Gemcitabine 1000mg Without Afatinib
Number analyzed (Participants) | 12 | 13
ng/mL | 16000.0 (32.1) | 13500.0 (43.8)
Statistical Analysis 1: Comparison: Gemcitabine 1000mg With Afatinib 40 mg vs Gemcitabine 1000mg Without Afatinib; Test type: Non-Inferiority or Equivalence — p-value for ratio outside interval 80% to 125%; p = 0.3359, ANOVA; [statistical method as in outcome 11, analysis 1]; Ratio of adjusted gmeans in percentage = 118.41, 90% CI 2-sided [94.81 to 147.88], Standard Deviation 31.6 — [estimate comment as in outcome 13, analysis 1]

15. Secondary Outcome: Total Clearance (CL) of Gemcitabine
Description: Total Clearance (CL) of Gemcitabine from plasma.
Time Frame: PK samples were taken on day 1 at hours; -0:05, 0:30, 1, 1:30, 2, 3 and on day 22 at hours; -0:10, 0:30, 1, 1:30, 2, 3
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Gemcitabine 1000mg With Afatinib 40 mg | Gemcitabine 1000mg Without Afatinib
Number analyzed (Participants) | 11 | 13
mL/min | 3020.0 (35.7) | 4090.0 (48.8)

16. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Gemcitabine
Description: Apparent volume of distribution at steady state (Vss) of Gemcitabine.
Time Frame: PK samples were taken on day 1 at hours; -0:05, 0:30, 1, 1:30, 2, 3 and on day 22 at hours; -0:10, 0:30, 1, 1:30, 2, 3
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Gemcitabine 1000mg With Afatinib 40 mg | Gemcitabine 1000mg Without Afatinib
Number analyzed (Participants) | 11 | 13
L | 90.5 (41.5) | 106.0 (59.8)

17. Secondary Outcome: AUC 0-24 of Docetaxel
Description: Area under the concentration-time curve of docetaxel in plasma over the time interval from 0 up to 24 hours
Time Frame: PK samples were taken on day 1 at hours; -0:05, 1, 2, 3, 5, 7, 23:55 and on day 22 at hours; -0:10, 1, 2, 3, 5, 7, 23:55
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Docetaxel 60mg With Afatinib 30mg: Afatinib (film-coated tablet) 30 mg qd (once daily) was administered orally in combination with Docetaxel 60 mg/m2 administered as intravenous infusion on Day 1 of each 3- week treatment course.
- Docetaxel 60mg Without Afatinib: Docetaxel 60 mg/m2 administered as intravenous infusion on Day 1 of each 3- week treatment course.
- Docetaxel 75mg With Afatinib 30mg: Afatinib (film-coated tablet) 30 mg qd (once daily) was administered orally in combination with Docetaxel 75 mg/m2 administered as intravenous infusion on Day 1 of each 3- week treatment course.
- Docetaxel 75mg Without Afatinib: Docetaxel 75 mg/m2 administered as intravenous infusion on Day 1 of each 3- week treatment course.
Arm/Group | Docetaxel 60mg With Afatinib 30mg | Docetaxel 60mg Without Afatinib | Docetaxel 75mg With Afatinib 30mg | Docetaxel 75mg Without Afatinib
Number analyzed (Participants) | 15 | 12 | 18 | 15
ng*h/mL | 2000.0 (41.4) | 2210.0 (41.7) | 2400.0 (50.9) | 2270.0 (46.4)
Statistical Analysis 1: Comparison: Docetaxel 60mg With Afatinib 30mg vs Docetaxel 60mg Without Afatinib; Test type: Non-Inferiority or Equivalence — p-value for ratio outside interval 80% to 125%; p = 0.0349, ANOVA; [statistical method as in outcome 11, analysis 1]; Ratio of adjusted gmeans in percentage = 93.69, 90% CI 2-sided [81.352 to 107.890], Standard Deviation 19.5 — Relative bioavailability of Docetaxel with Afatinib vs. Docetaxel without Afatinib was estimated by the ratios of the adjusted geometric means (gMean). Standard deviation is actually intra-individual geometric coefficient variation (gCV)
Statistical Analysis 2: Comparison: Docetaxel 75mg With Afatinib 30mg vs Docetaxel 75mg Without Afatinib; Test type: Non-Inferiority or Equivalence — p-value for ratio outside interval 80% to 125%; p = 0.0405, ANOVA; [statistical method as in outcome 11, analysis 1]; Ratio of adjusted gmeans in percentage = 98.11, 90% CI 2-sided [81.053 to 118.760], Standard Deviation 30.4 — [estimate comment as in outcome 17, analysis 1]

18. Secondary Outcome: Cmax of Docetaxel
Description: Maximum concentration of docetaxel in plasma.
Time Frame: as for outcome 17
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Docetaxel 60mg With Afatinib 30mg | Docetaxel 60mg Without Afatinib | Docetaxel 75mg With Afatinib 30mg | Docetaxel 75mg Without Afatinib
Number analyzed (Participants) | 15 | 15 | 18 | 18
ng/mL | 1690.0 (42.8) | 1860.0 (36.0) | 1790.0 (61.7) | 2080.0 (60.0)
Statistical Analysis 1: Comparison: Docetaxel 60mg With Afatinib 30mg vs Docetaxel 60mg Without Afatinib; Test type: Non-Inferiority or Equivalence — p-value for ratio outside interval 80% to 125%; p = 0.0728, ANOVA; [statistical method as in outcome 11, analysis 1]; Ratio of adjusted gmeans in percentage = 90.78, 90% CI 2-sided [78.566 to 104.901], Standard Deviation 22.8 — [estimate comment as in outcome 17, analysis 1]
Statistical Analysis 2: Comparison: Docetaxel 75mg With Afatinib 30mg vs Docetaxel 75mg Without Afatinib; Test type: Non-Inferiority or Equivalence — p-value for ratio outside interval 80% to 125%; p = 0.3294, ANOVA; [statistical method as in outcome 11, analysis 1]; Ratio of adjusted gmeans in percentage = 85.74, 90% CI 2-sided [65.561 to 112.138], Standard Deviation 48.9 — [estimate comment as in outcome 17, analysis 1]

19. Secondary Outcome: Total Clearance (CL) of Docetaxel
Description: Total Clearance (CL) of Docetaxel from plasma.
Time Frame: as for outcome 17
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Docetaxel 60mg With Afatinib 30mg | Docetaxel 60mg Without Afatinib | Docetaxel 75mg With Afatinib 30mg | Docetaxel 75mg Without Afatinib
Number analyzed (Participants) | 14 | 12 | 14 | 15
mL/min | 811.0 (38.0) | 671.0 (47.6) | 886.0 (34.7) | 892.0 (49.5)

20. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Docetaxel
Description: Apparent volume of distribution at steady state (Vss) of Docetaxel.
Time Frame: as for outcome 17
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Docetaxel 60mg With Afatinib 30mg | Docetaxel 60mg Without Afatinib | Docetaxel 75mg With Afatinib 30mg | Docetaxel 75mg Without Afatinib
Number analyzed (Participants) | 14 | 12 | 14 | 15
L | 255.0 (73.9) | 315.0 (56.9) | 323.0 (66.2) | 300.0 (68.9)

ADVERSE EVENTS:
Time Frame: From first drug administration until 28 days after last drug administration, up to 717 days
Arm/Group | Afatinib 30mg and Gemcitabine 1000mg | Afatinib 30mg and Gemcitabine 1250mg | Afatinib 40mg and Gemcitabine 1000mg | Afatinib 40mg and Gemcitabine 1250mg | Afatinib 50mg and Gemcitabine 1250mg | Afatinib 30mg and Docetaxel 60mg | Afatinib 30mg and Docetaxel 75mg | Afatinib 40mg and Docetaxel 75mg | Afatinib 50mg and Docetaxel 75mg
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/8 | 12/20 | 2/6 | 2/2 | 7/18 | 15/18 | 8/12 | 6/6
Other Adverse Events (participants affected / at risk) | 3/3 | 8/8 | 20/20 | 6/6 | 2/2 | 18/18 | 18/18 | 12/12 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 30mg and Gemcitabine 1000mg (N=3) | Afatinib 30mg and Gemcitabine 1250mg (N=8) | Afatinib 40mg and Gemcitabine 1000mg (N=20) | Afatinib 40mg and Gemcitabine 1250mg (N=6) | Afatinib 50mg and Gemcitabine 1250mg (N=2) | Afatinib 30mg and Docetaxel 60mg (N=18) | Afatinib 30mg and Docetaxel 75mg (N=18) | Afatinib 40mg and Docetaxel 75mg (N=12) | Afatinib 50mg and Docetaxel 75mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 4 | 1 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Performance status decreased (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis syndrome (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sphingomonas paucimobilis infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 0 | 0 | 1 | 2 | 1 | 2
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelocaliectasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Ureteric stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 30mg and Gemcitabine 1000mg (N=3) | Afatinib 30mg and Gemcitabine 1250mg (N=8) | Afatinib 40mg and Gemcitabine 1000mg (N=20) | Afatinib 40mg and Gemcitabine 1250mg (N=6) | Afatinib 50mg and Gemcitabine 1250mg (N=2) | Afatinib 30mg and Docetaxel 60mg (N=18) | Afatinib 30mg and Docetaxel 75mg (N=18) | Afatinib 40mg and Docetaxel 75mg (N=12) | Afatinib 50mg and Docetaxel 75mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 12 | 2 | 0 | 5 | 11 | 4 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 3 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 7 | 2 | 0 | 9 | 14 | 7 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 3 | 0 | 0 | 1 | 3 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1
Ichthyosis (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eyelid irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 3 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Xerophthalmia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 4 | 0 | 0 | 5 | 1 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 1 | 1 | 3 | 2 | 2
Abdominal rigidity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aerophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anal inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 6 | 1 | 2 | 7 | 3 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 7 | 16 | 5 | 1 | 14 | 17 | 12 | 4
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 4 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 12 | 3 | 2 | 7 | 6 | 5 | 4
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral mucosal eruption (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Reflux gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 3 | 9 | 5 | 1 | 13 | 13 | 7 | 4
Vomiting (Gastrointestinal disorders) | 1 | 2 | 10 | 3 | 1 | 10 | 6 | 3 | 4
Asthenia (General disorders) | 1 | 5 | 14 | 3 | 2 | 14 | 11 | 8 | 5
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 2 | 1
Chills (General disorders) | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 6 | 1 | 0 | 2 | 3 | 2 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Localised oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 1 | 3 | 0 | 0 | 2 | 1 | 2 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 2 | 3 | 2 | 0 | 4 | 5 | 2 | 1
Pain (General disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 2 | 5 | 0 | 0 | 7 | 5 | 4 | 1
Ulcer (General disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1 | 2 | 2 | 1 | 1 | 2 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bursitis infective staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 3 | 0 | 0 | 1 | 4 | 1 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1
Gastrointestinal fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Genital infection fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 1 | 2 | 9 | 1 | 0 | 5 | 6 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pleural infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 4 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Superinfection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 3 | 1
Urinary tract infection staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vulvitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Burn oesophageal (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Face crushing (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 3 | 4 | 1 | 0 | 2 | 1 | 0 | 0
Aortic bruit (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 3 | 5 | 1 | 0 | 1 | 1 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Blood iron decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Blood urea increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Epidermal growth factor receptor decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 2 | 1 | 0 | 1 | 2 | 1 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 2 | 0 | 8 | 3 | 0 | 3 | 7 | 4 | 4
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 4 | 10 | 3 | 2 | 9 | 8 | 8 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Feeding disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 0 | 4 | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 3 | 1 | 2 | 1 | 2 | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 5 | 2 | 0 | 3 | 3 | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 1 | 0 | 2 | 5 | 2 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypouricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 3 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 0 | 0 | 2 | 1 | 3 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2 | 0 | 2 | 4 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 2 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aphonia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 0 | 1 | 2 | 0 | 3 | 2 | 2 | 0
Headache (Nervous system disorders) | 1 | 2 | 4 | 0 | 0 | 5 | 1 | 3 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Motor dysfunction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 4 | 0 | 0 | 1 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 3 | 2 | 0 | 0 | 2 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 2
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital paraesthesia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Penile erythema (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Penile oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 6 | 2 | 0 | 3 | 2 | 4 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 5 | 1 | 0 | 5 | 3 | 3 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 5 | 2 | 0 | 5 | 5 | 6 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 0 | 3 | 2 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 4 | 4 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 4 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 4 | 8 | 1 | 0 | 4 | 8 | 7 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 1 | 0 | 2 | 0 | 2 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Mucocutaneous rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 5 | 12 | 4 | 1 | 6 | 13 | 6 | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 1 | 4 | 1 | 0 | 5 | 3 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 0
Skin oedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 1 | 1 | 2 | 1 | 0
Skin warm (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arterial thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.